CLINICAL TRIAL: NCT01272752
Title: Surveillance Study of Weight Response and Body Composition in Subjects Who Are First-Time Users (Less Than 3 Months) of the Following Medications: Risperdal, Seroquel, and/or Zyprexa, in Combination With 500 mg IHBG-10 TID
Brief Title: Anti-psychotic Medication (New Use) Weight Loss Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study did not get started.
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARI-1310-IHBG10
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Obesity
Keywords: obesity; weight loss; weight management; anti-psychotic medication; nutriceutical
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study Group (Experimental): Subjects will take 500 mg IHBG-10 15 minutes prior to the three main meals of the day.
  Interventions: Dietary Supplement: IHBG-10
- Control Group (Placebo Comparator): Subjects will take a placebo 15 minutes prior to the three main meals of the day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: IHBG-10 — 500 mg IHBG-10
  Other Names: IHBG10
  Arms: Study Group
Dietary Supplement: Placebo — Placebo taken 15 minutes prior to the three main meals of the day
  Other Names: sugar pill
  Arms: Control Group

SUMMARY:
This is a pilot study to determine the safety and efficacy of an investigational product (IHBG-10) on weight change and changes in body composition in subjects who have just started taking (for less than three months) certain anti-psychotic medications (Risperdal, Seroquel, and/or Zyprexa).

DETAILED DESCRIPTION:
A total of 30 subjects will be enrolled in this study. They will be randomized in to one of two groups. One group (of 20 subjects) will take 500 mg of the investigational product (IHBG-10) 15 minutes prior to the three main meals of the day; subjects will continue to take their prescribed anti-psychotic medications. The other group (of 10 subjects) will take a placebo 15 minutes prior to the three main meals of the day; subjects will continue to take their prescribed anti-psychotic medications. Subjects will take the investigational product or placebo for 12 weeks. Participation in this study involves 4 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 and older
* Agree to keep diet, exercise and all current health habits stable during participation in the study
* Have been taking Risperdal (Risperidone), Seroquel (Quetiapine), or Zyprexa (Olanzapine) for less than 3 months

Exclusion Criteria:

* Current active acute psychotic episode
* Women who are pregnant, breastfeeding or planning to become pregnant
* Prior bariatric surgery
* Use of prescription or over-the-counter appetite suppressants, herbal products or other medications for weight loss within the past month
* Obesity as a result of a clinically-diagnosed endocrine problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Weight | 12 weeks

SECONDARY OUTCOMES:
Body composition | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Soundy, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Research Institute, Sioux Falls, South Dakota, United States